CLINICAL TRIAL: NCT04155619
Title: Using Early Time Restricted Feeding and Timed Light Therapy to Improve Glycemic Control in Adults With Type 2 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Courtney M Peterson, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300003964; W81XWH-19-1-0558 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2; Time Restricted Feeding; Light; Therapy, Complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Intermittent Fasting | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The study statistician will be blinded. To the degree possible for each task, other study staff will be blinded during outcome assessments and analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No change in eating or light exposure habits (Active Comparator)
  Interventions: Behavioral: No change in meal timing; Behavioral: No change in light exposure
- Early Time-Restricted Feeding (Experimental)
  Interventions: Behavioral: No change in light exposure; Behavioral: Early Time-Restricted Feeding
- Timed Light Therapy (Experimental)
  Interventions: Behavioral: No change in meal timing; Behavioral: Timed Light Therapy
- Early Time-Restricted Feeding and Timed Light Therapy (Experimental)
  Interventions: Behavioral: Early Time-Restricted Feeding; Behavioral: Timed Light Therapy

INTERVENTIONS:
Behavioral: No change in meal timing — Participants will eat within an ≥11-hour daily period (no change in meal timing habits).
  Arms: No change in eating or light exposure habits; Timed Light Therapy
Behavioral: No change in light exposure — Participants will not change their light exposure habits.
  Arms: Early Time-Restricted Feeding; No change in eating or light exposure habits
Behavioral: Early Time-Restricted Feeding — Participants will eat within an 8-hour daily period early in the day, starting within 2 hours of waking up.
  Other Names: eTRF, early TRF
  Arms: Early Time-Restricted Feeding; Early Time-Restricted Feeding and Timed Light Therapy
Behavioral: Timed Light Therapy — Participants will use bright light therapy for 60 minutes between 6 am - 3 pm, blue light-blocking glasses for one hour before bedtime, and blackout curtains at night.
  Other Names: Bright Light Therapy
  Arms: Early Time-Restricted Feeding and Timed Light Therapy; Timed Light Therapy

SUMMARY:
The purpose of this study is to test whether eating earlier in the day and/or timed light therapy can improve blood sugar in people with type 2 diabetes. This study will also test whether these treatments improve other aspects of health, including the circadian (biological) clock, sleep, weight, body composition, cardiovascular health, quality of life, and mood.

DETAILED DESCRIPTION:
The circadian system is strongly linked to type 2 diabetes. Adults with type 2 diabetes have circadian rhythms that are both weakened and mistimed. Weak rhythms may be due to insufficient bright light exposure during the daytime, irregular meal timing, or grazing on food throughout the day. Mistiming may be due to ill-timed food intake or light exposure-such as eating later in the day or light exposure at night-which causes central and peripheral circadian clocks within the body to become out of sync (circadian misalignment). This circadian misalignment impairs glucose metabolism: data now show that eating late in the day and light exposure at night rapidly elevate glucose (blood sugar) and insulin levels in humans within days. Conversely, well-timed food intake and light exposure appear to improve glycemic (blood sugar) control, circadian rhythms, and several other aspects of health.

This study will test the health effects of eating early in the daytime (early time-restricted feeding; early TRF) and timed light therapy in adults with type 2 diabetes. The study will test the following aims:

1. Determine whether early TRF and/or timed light therapy improve glycemic control
2. (a) Determine how early TRF and/or timed light therapy affect the central and peripheral circadian clocks and (b) determine which patients benefit the most from circadian-based therapies
3. Determine whether early TRF and/or timed light therapy improve sleep, body weight, body composition, cardiovascular risk factors, quality of life, and psychological health.

Approximately 344 veterans and civilians aged 30-80 with insulin-independent type 2 diabetes will be randomized to the following 2 x 2 study design:

1. No change in eating or light exposure habits
2. Early TRF
3. Timed light therapy
4. Early TRF and timed light therapy

Participants will be asked to follow their assigned treatment for 16 weeks and then be followed up for an additional eight months (1 year in total). Baseline and post-intervention testing will be conducted during a 38-hour inpatient (hospital) stay. Testing will involve three 3-hour meal tolerance tests to determine insulin sensitivity and secretion; 24-hour measurement of glucose, insulin, and C-peptide levels; 24-hour measurement of cortisol and melatonin to measure the phase and amplitude of the central clock; and a constant glucose infusion to determine the phase and amplitude of the effective glycemic ("peripheral") circadian clock. Sleep, weight loss, body composition, and cardiovascular risk factors will also be measured, and questionnaires and an interview will be administered to determine improvements in quality of life and psychological health.

Note: Pre-registered primary and secondary outcomes are listed below. Pre-registered tertiary outcomes appear in the study protocol, which will be uploaded to this website.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-80 years old
* Have type 2 diabetes
* HbA1c between 5.7 - 12.0%
* On a stable dose of metformin, DPP-IV inhibitors, SGLT2 inhibitors, sulfonylureas, and/or GLP-1 receptor agonists for at least 6 weeks, or taking no diabetes medications
* Wake up at a regular time between 5-9 am

Exclusion Criteria:

* On insulin or diabetes medication other than metformin, DPP-IV inhibitors, SGLT2 inhibitors, sulfonylureas, and/or GLP-1 receptor agonists
* Have type 1 diabetes or was diagnosed with diabetes before age 18
* Moderate or severe retinopathy or other medical condition that may affect the ability to safely receive bright light therapy
* A history of severe hypoglycemia
* Change in the dosage of a chronic medication within the past month (need to wait at least 1 month prior to baseline visit)
* Have a clinically significant laboratory abnormality (e.g., abnormal hemoglobin levels)
* Severe gastrointestinal disease, major gastrointestinal surgery, or active gallstone disease
* Cardiovascular, renal, cardiac, liver, lung, adrenal, or nervous system disease that is unstable or may compromise study validity
* Evidence of cancer (other than non-melanoma skin cancer) within the last 5 years
* Pregnant or breastfeeding
* Current diagnosis of a major psychiatric condition that would impair study participation
* Diagnosed sleep disorder or circadian disorder that is not stabilized (sleep apnea is allowed). Those with narcolepsy will not be included.
* Major changes in health or medical history in the last 3 months that could affect data validity per judgement of the study physician
* Spend an average of more than 1.5 hours/day outdoors
* Perform overnight shift work more than 1 day/week on average
* Regularly eat within a less than a 10-hour period daily
* Regularly finish eating dinner before 6:30 pm
* Lost or gained more than 8 lbs within the last 2 months and weight needs to be stable for a minimum of 4 weeks before baseline testing
* Traveled more than two times zones away in the two months prior to enrolling in the trial or will travel more than two time zones away during the 16-week study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
24-hour glucose levels | 16 weeks
  Time-weighted mean, fasting, peak, standard deviation, and excursion (maximum - minimum) values (mg/dl)
24-hour insulin levels | 16 weeks
  Time-weighted mean, fasting, peak, standard deviation, and excursion values (mU/l)
24-hour C-peptide levels | 16 weeks
  Time-weighted mean, fasting, peak, standard deviation, and excursion values (pmol/l). This is also a proxy for total 24-hour insulin secretion.
Hemoglobin A1C | 16 weeks
  %
Insulin sensitivity | 16 weeks
  Insulin sensitivity (dl/kg/min/μU/ml) during three identical meal tolerance tests, as measured by the Oral Minimal Model. The individual, mean, and excursion values, and time of the peak value will also be calculated.
Beta-cell responsivity index (a measure of beta-cell function) | 16 weeks
  Beta-cell responsivity during three identical meal tolerance tests, as measured by the Oral Minimal Model. The individual, mean, and excursion values, and time of the peak value will also be calculated.
Insulin secretion | 16 weeks
  Insulin secretion (mU) across three identical meal tolerance tests, as measured by the Oral Minimal Model. The individual, mean, and excursion values, and time of the peak value will also be calculated.

SECONDARY OUTCOMES:
Melatonin Amplitude | 16 weeks
  Peak value (pg/mL)
Cortisol Amplitude | 16 weeks
  Amplitude (μg/dl)
Melatonin Phase | 16 weeks
  Clock time of dim light melatonin onset (DLMO)
Cortisol Phase | 16 weeks
  Clock time of cortisol phase
Glycemic ("Peripheral") Rhythm Amplitude | 16 weeks
  Amplitude or diurnal variation in glucose levels (mg/dl) during a constant glucose infusion procedure
Glycemic ("Peripheral") Rhythm Phase | 16 weeks
  Time of day that glucose levels experience a nadir during a constant glucose infusion procedure

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Peterson, Ph.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham; Birmingham Veterans Affairs Medical Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes